CLINICAL TRIAL: NCT06349460
Title: A Micro-Randomized Trial to Optimize Just-in-Time Adaptive Intervention for Binge Eating & Weight-related Behaviors
Brief Title: Trial to Optimize Just-in-Time Adaptive Intervention for Binge Eating & Weight-related Behaviors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Graham, Associate Professor, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00216998; R01DK133300 (NIH)
Record Dates: First submitted 2024-03-30; First posted 2024-04-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Binge Eating; Obesity
MeSH Terms: conditions — Bulimia; Obesity

STUDY DESIGN:
Intervention Model Description: In this micro-randomized trial, participants will have 2 consecutive, independent micro-randomizations at the time of target selection each week for 16 weeks: namely, 1 of 5 treatment targets will be randomly delivered, either as a recommended or assigned target, to each user, of equal probability per randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Increase healthy eating behaviors - Assigned (Experimental): Individuals will be assigned to increase healthy eating behaviors that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Increase healthy eating behaviors - Recommended (Experimental): Individuals will be recommend to increase healthy eating behaviors that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Increase physical activity - Assigned (Experimental): Individuals will be assigned to increase physical activity that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Increase physical activity - Recommended (Experimental): Individuals will be recommended to increase physical activity that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Limit unhealthy dieting behaviors - Assigned (Experimental): Individuals will be assigned to limit unhealthy dieting behaviors that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Limit unhealthy dieting behaviors - Recommended (Experimental): Individuals will be recommended to limit unhealthy dieting behaviors that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Improve self-image - Assigned (Experimental): Individuals will be assigned to improve self-image that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Improve self-image - Recommended (Experimental): Individuals will be recommended to improve self-image that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Improve mood - Assigned (Experimental): Individuals will be assigned to improve mood that week.
  Interventions: Behavioral: FoodSteps behavioral intervention
- Improve mood - Recommended (Experimental): Individuals will be recommended to improve mood that week.
  Interventions: Behavioral: FoodSteps behavioral intervention

INTERVENTIONS:
Behavioral: FoodSteps behavioral intervention — Behavioral intervention that targets binge eating and weight-related behaviors. Each week, users are recommended or assigned one of five targets, set a relevant goal, and track their progress. If a target is recommended, the user can choose to select that target or a different target.

SUMMARY:
The purpose of this study is to conduct a micro-randomized trial to learn which evidence-based targets within a mobile intervention for binge eating and weight-related behaviors are most impactful for which people and in what sequence.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Obesity (BMI ≥30)
* Recurrent binge eating (≥12 episodes in the past 3 months)
* Interested in losing weight and reducing binge eating
* Willing to use a mobile application
* Has a smartphone with Internet access and capacity for calls and text messaging
* Has a valid email address
* Has access to a scale
* Not pregnant
* English-speaking

Exclusion Criteria:

* Diagnosis for which the study/intervention is not clinically indicated
* Not currently receiving clinical services for weight management or binge eating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weekly change in binge eating | 1 week
  Change in number of binge eating episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ortega A, Rooper IR, Massion T, Azubuike C, Lipman LD, Lakhtakia T, Camino MK, Parsons LM, Tack E, Alshurafa N, Kay M, Graham AK. Co-designing prediction data visualizations for a digital binge eating intervention. Transl Behav Med. 2025 Jan 16;15(1):ibaf009. doi: 10.1093/tbm/ibaf009. PMID 40167045